CLINICAL TRIAL: NCT00555139
Title: Double-blind, Randomized, Placebo and Alprazolam-controlled Three-period Crossover Incomplete Block Design Study to Compare Putative Anxiolytic-like fRMI Activity of GW876008 and GSK561679 After Single-dose Administration in Subjects With Social Anxiety Disorder (SAD)
Brief Title: A Study To Compare The Putative Anxiolytic Effect Of 2 New Drugs In Subjects With Social Anxiety Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: CRH108571
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Social Phobia
Keywords: anxiety,; depression,; fMRI; CRF-1 antagonists,
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders; Depression | interventions — NBI 77860; GW 876008; Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW876008 (Experimental): The subjects will be randomized to one of the six sequences A/B/D A/D/B B/A/D B/D/A D/A/B D/B/A across three treatment periods where A represents placebo, B represents GW876008 and D represents alprazolam.
  Interventions: Drug: GW876008 tablet; Drug: alprazolam; Drug: Placebo
- GSK561679 (Experimental): The subjects will be randomized to one of the six sequences A/C/D A/D/C C/A/D C/D/A D/A/C D/C/A across three treatment periods where A represents placebo, C represents GSK561679 and D represents alprazolam.
  Interventions: Drug: GSK561679 tablet; Drug: alprazolam; Drug: Placebo

INTERVENTIONS:
Drug: GSK561679 tablet — GSK561679 tablets are white film-coated tablets, containing 200 (milligrams) mg of the free base, GSK561679A.
  Arms: GSK561679
Drug: GW876008 tablet — GW876008 tablets are white to off-white round film-coated tablets, containing 100 mg of GW876008X (free base).
  Arms: GW876008
Drug: alprazolam — Alprazolam capsules 0.25 mg are hard gelatine capsules containing 1 tablet of commercial alprazolam (Xanax 0.25).
  Other Names: GSK561679; GW876008
Drug: Placebo — GW876008 placebo tablets will visually match the active GW876008 tablets. GSK561679 placebo tablets will visually match the active GSK561679 tablets. Placebo to match Alprazolam is a hard gelatine capsule that will visually match the active but containing only a filler.

SUMMARY:
To compare by neuroimaging techniques and public speaking, the way social anxiety patients respond after the administration of GW876008, GSK561679, alprazolam and placebo

ELIGIBILITY:
Inclusion criteria:

* Outpatient with a primary diagnosis of Social Anxiety
* LSAS score of 50 or more.
* Men or women who are between 18 and 64 years of age. Women will be included in this study only if the reproductive toxicology data available at the time of study start will allow their inclusion, in accordance with regulatory requirements.
* Body weight > 50 kg and BMI within the range 18.5 - 31.0 kg/m2.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject must be able to read, comprehend and record information.
* A signed and dated written informed consent is obtained from the subject.
* Subjects willing to restrict alcohol intake to 4 unit of alcohol or less per day. A unit is equivalent to 300 ml of beer or one measure of spirits or one glass of wine.
* Women must be of non child bearing potential or commit to consistent and correct use of an acceptable method of birth control that must be recorded on the source documentation at screening and verified for continued compliance at each visit; GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of a physician, are as follows:
* Subjects with a history of peptic ulcer disease (PUD) with a known aetiology must provide documentation by a gastroenterologist of the aetiology of the PUD and that effective treatment was provided with full eradication of ulcers and symptoms.

Exclusion criteria:

* Any concomitant drug dosing 24 h before each dosing.
* Any history of a clinically significant abnormality of the neurological system (including dementia and other cognitive disorders or significant head injury) or any history of seizure (excluding febrile seizure).
* Subjects with an unstable medical disorder or a disorder that would likely interfere with the action, absorption, distribution, metabolism or excretion of GW876008, GSK561679 or alprazolam, may pose a safety concern, or interfere with accurate assessment of safety.
* The subject has a current or recent (within six months) documented gastrointestinal disease
* Subject has symptoms of the presenting illness which are better accounted for by another diagnosis or subjects who meet DSM-IV criteria for any other Axis I disorder as a primary diagnosis currently or within 6 months prior to the screening visit or A current DSM-IV-TR diagnosis of Antisocial or Borderline Personality Disorder, Dementia, or another current DSM-IV-TR Axis II diagnosis that would suggest nonresponsiveness to pharmacotherapy or non-compliance with the protocol; or A current (or within six months prior to the Screening visit) diagnosis of anorexia nervosa or bulimia; or Subjects with a history of Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder.
* HAMD-17 score greater than 15.
* Subjects who are currently receiving regularly scheduled psychotherapy (individual or group, including cognitive behavioural therapy), plan to initiate psychotherapy during the trial or have received regularly scheduled psychotherapy during the 12 week period prior to the Screening Visit.
* Subjects have any laboratory abnormality that in the investigator's judgment is considered to be clinically significant and not resolved by the Randomization Visit.
* The subject has a semi-supine systolic blood pressure less than 90mmHg (85mmHg for females) or greater than 140mmHg or a semi-supine diastolic blood pressure of less than 45mmHg or greater than 90mmHg; or a pulse rate less than 40bpm or more than 90bpm.
* Women who have a positive serum Human Chorionic Gonadotropin (HCG) pregnancy test at screen visit, a positive urine dipstick test at Randomization, or who are lactating or planning to become pregnant within the next 2weeks after the Follow Up Visit.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 60 days or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* As a result of any of the medical interview, physical examination or screening investigations the physician responsible considers the subject unfit for the study.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John'sWort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety
* Subjects who, in the opinion of the investigator, would be noncompliant with the visit schedule or study procedures (e.g., illiteracy, planned vacations, or planned hospitalizations during the study).
* Subjects who are not euthyroid as evidenced by normal TSH. Subjects maintained with thyroid medication must be euthyroid for a period of at least six months prior to the screen visit.
* Subject's level of FSH falling outside normal range
* Subjects with diabetes or high risk of diabetes based on a documented history of impaired glucose tolerance.
* Subjects have any electrocardiographic (ECG) parameter outside of the Sponsor-specified ranges at either screen or randomization visit.
* Subjects who have had electroconvulsive therapy (ECT) or transcranial magnetic stimulation within the 6 months prior to the Screening Visit.
* Subjects, who are left-handed.
* The subject has a positive pre-study urine drug/ breath alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Documented history of hepato-biliary disease or abnormality in hepatic enzymesat screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2007-03-27 (Actual); Primary Completion 2008-01-10 (Actual); Study Completion 2008-01-10 (Actual)

PRIMARY OUTCOMES:
Changes of fMRI activation in amygdala of subjects with SAD during an emotional task after having received different compounds. Change in the VAS score in response to Public Speaking stress after having received different compounds. | over 6 weeks

SECONDARY OUTCOMES:
Changes of fMRI activation patterns in all brain areas in subjects with SAD during an emotional task or resting state. Changes of cortisol levels and other stress indicators in response to Public Speaking stress. | over 6 weeks
Pk samples: | 2 hours,4-5, 8hours post-dose (over 3 weeks, week 1,2&3)
Cortisol, ACTH: | 5hours 20min,5hours 35 min, 6hours & 7hours post dose (over 6 weeks, week 1,2,3 &6)
Indicators of physiological state during the fMRI session: | pre-dose, 5hours 20mins, 5hours 43mins, 6 hours, 6hours 20mins (over 6 weeks, week 1,2,3 &6)
Heart rate (HR), Respiratory rate (RR), ventilation (pneumatic pletismography), and carbon dioxide percutaneous measurements monitored during the whole procedure (control and exploratory profile tests). | pre-dose, 5hours 20mins, 5hours 43mins, 6 hours, 6hours 20mins (over 6 weeks, week 1,2,3 &6)
Visual Analog Scale (VAS) measurements of distress | 3.5-4hours, 4.5-5.3hours, 5hours 20mins, 5hours 35mins, 5hours 43mins after public speaking, 6hours, 6hours 20mins, 7hours (week 1,2, and 3)
Maddox wing test. | Week 1, 2 and 3
questionnaire for sédation. | Week 1, 2 and 3
plasma levels of the various compounds to derive pharmacokinetic parameters | 1hour, 2hours, 4-5hours, 8hours (week 1, 2 and 3)
Safety and tolerability will be evaluated by adverse event monitoring, physical examination, ECG, vital signs and laboratory parameters | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Mataro (Barcelona)
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Terrassa - Barcelona

REFERENCES:
- See also: Results for study CRH108571 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CRH108571?search=study&search_terms=CRH108571#rs